CLINICAL TRIAL: NCT04861870
Title: Bandebereho Randomized Control Trial: Six Year Follow-up to Assess the Impact of a Gender-transformative Intervention With Couples to Promote Men's Engagement in Maternal, Newborn and Child Health, Caregiving and Healthier Couple Relations
Brief Title: Bandebereho 6 Year Follow up RCT in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Promundo, United States (Other)
Collaborators: Rwanda Men's Resource Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RWN6YR
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Gender Relations; Violence; Child Development; Contraception; Prenatal Care; Partner Communication
Keywords: Gender; Violence; Early childhood development (ECD); Caregiving; Parenting; MNCH; Reproductive health
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): See intervention description
  Interventions: Behavioral: MenCare+/Bandebereho fathers'/couples' group education
- Control (No Intervention): Participants randomized into the control arm are surveyed at the same time points as intervention participants, but did not receive any intervention.

INTERVENTIONS:
Behavioral: MenCare+/Bandebereho fathers'/couples' group education — MenCare+/Bandebereho was a 3 year project to engage men in maternal, newborn and child health (MNCH) and in sexual and reproductive health in Rwanda. A core component of the project is fathers'/couples' group education. The target participants were first-time parents or parents of young children living in 16 rural and semi-urban sectors selected by the implementing partner in collaboration with local authorities. The MenCare+/Bandebereho fathers'/couples' group education engaged men in 15 weekly sessions of group discussion, critical reflection and interactive activities led by a trained facilitator using a curriculum developed by RWAMREC and Promundo and approved by the Rwandan Ministry of Health, adapted from the Program P Manual. Men's partners participate in 6-8 sessions. The sessions focused on men's role in MNCH, family planning, sharing household responsibilities, intimate partner violence, conflict resolution, family budgeting, and gender equality.
  Other Names: Program P
  Arms: Intervention

SUMMARY:
This study seeks to conduct a six-year follow-up of the Bandebereho randomized control trial (RCT) to assess the longer-term impact of the gender-transformative Bandebereho couples intervention on participating men, women, and their children. The Bandebereho program was implemented by the Rwanda Men's Resource Centre (RWAMREC) and Promundo-US, in collaboration with the Rwanda Ministry of Health and local authorities between 2013 and 2015. A two-arm RCT collected three rounds of data from 1,199 couples (575 treatment; 624 control) starting in 2015-16: baseline (pre-intervention), 9 month follow-up, and 21-month follow-up. The findings at 21-months demonstrated significant impacts of the intervention on multiple gender and health-related outcomes. This study will conduct surveys with men enrolled in the RCT and their female partners 6 years after the intervention, to assess its long-term impact on reproductive and maternal health, gender attitudes and household dynamics, intimate partner violence, mental health and wellbeing, parenting, and child development. In addition, child assessments will be conducted with a sub-sample of 800 children aged 4 to 7 years to directly assess early childhood development outcomes.

DETAILED DESCRIPTION:
This study seeks to conduct a six-year follow-up of the Bandebereho randomized controlled trial (RCT) to assess the longer-term impact of the gender-transformative Bandebereho couples intervention on participating men, women, and their children. The Bandebereho program being assessed was first implemented by the Rwanda Men's Resource Center (RWAMREC) and Promundo-US, in collaboration with the Rwanda Ministry of Health and local authorities in Karongi, Musanze, Nyaruguru and Nyaruguru districts between 2013 and 2015. A two-arm RCT was conducted with 1,199 couples (575 treatment; 624 control) in 2015-16. Three rounds of data were collected: baseline (pre-intervention), 9 month follow-up (4 months post-intervention), and 21-month follow-up (16 months post-intervention). The findings at 21-months demonstrated significant impacts of the intervention on multiple gender and health-related outcomes. The proposed study will conduct surveys with men enrolled in the RCT and their female partners, to assess the longer-term impact of the intervention on reproductive and maternal health, gender attitudes and household dynamics, intimate partner violence, mental health and wellbeing, parenting, and child development. In addition, child assessments will be conducted with a sub-sample of 800 children aged 4 to 7 years to directly assess early childhood development outcomes.

ELIGIBILITY:
Inclusion Criteria at baseline:

* Men aged 21-35 years
* Living with a partner
* Expectant (or soon to be) father or father of young children under-5
* Living in an area with a group facilitator

Exclusion Criteria at baseline:

- Participated in previous cycles of the same intervention

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 2818 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Women's experiences of intimate partner violence (physical & sexual) | Experience of violence in past 12 months, measured 6 years post intervention
  A composite capturing self-reported exposure to a standard set of violent acts by a partner in past 12 months, adapted from World Health Organisation's multi-country study on violence against women.
Use of violence/harsh punishment against children | 6 years post intervention
  A composite capturing respondents' self reported use of various harsh discipline acts in the past month, adapted from the UNICEF Multiple Indicator Cluster Surveys (MICS) study.
Observation-based child development measure | 6 years post intervention
  Observation-based scores on the International Development and Early Learning Assessment (IDELA) for children ages 4-7
Child behavior assessment | 6 years post intervention
  Parent-reported scores on Strengths and Difficulties Questionnaire (SDQ)

SECONDARY OUTCOMES:
Family planning | 6 years post intervention
  Self reported responses on current use of family planning methods, using Demographic and Health Survey (DHS) measure.
Antenatal care (ANC) service utilization | 6 years post intervention
  Self reported responses on women's frequency of ANC visits during most recent pregnancy, using DHS measure (women only).
Antenatal care (ANC) accompaniment | 6 years post intervention
  Self reported responses on men's frequency of accompaniment to ANC visits during most recent pregnancy, adapted from International Men and Gender Equality Survey.
Parenting behaviors with children | 6 years post intervention
  Composite variable capturing behaviors with children in the past week (e.g. reading stories, playing, etc.) adapted from IDELA HOME and select items related to parenting behaviors adapted from the Parenting and Family Adjustment Scales (PAFAS).
Parenting behaviors and adjustment | 6 years post intervention
  Select items related to parenting behaviors and feelings adapted from the Parenting and Family Adjustment Scales (PAFAS).
Time spent/gender division of caregiving/domestic tasks and paid work | 6 years post intervention
  a) A composite measure of self-reported time spent on specific tasks in the past week; and b) self-reported distribution of tasks between partners.

OTHER OUTCOMES:
Couple communication | 6 years post intervention
  A composite capturing frequency of communication across multiple topics.
Gender-related attitudes | 6 years post intervention
  A continuous scale variable, adapted from the validated Gender Equitable Men (GEM) scale; scores range from 1 to 5, with higher scores indicating more equitable attitudes.
Decision-making in relationship | 6 years post intervention
  Self-reported responses on who makes the decision in the relationship, adapted from the DHS.
Frequency of quarreling | 6 years post intervention
  Self-reported response to one item capturing frequency of quarreling in the couple.
Relationship quality and conflict resolution | 6 years post intervention
  Self-reported relationship quality items adapted from the relationship quality scale from the Decision Making in Low-Income Couples scale.
Relationship conflict resolution | 6 years post intervention
  Self-reported items on couple communication and resolution in conflict adapted from the Couple Functionality Assessment.
Alcohol use | 6 years post intervention
  Self reported alcohol use (men & women) and women's reports on partners' alcohol use (women) in past year, adapted from the Alcohol Use Disorders Identification Test (AUDIT).
Depression/Mental health | 6 years post intervention
  Self reported symptoms in past week, adapted from the Center for Epidemiologic Studies Depression Scale (CES-D) short form.
Reproductive coercion | Coercion in the past year, measured 6 years post intervention
  Women's self reported experience with reproductive coercion from their current partner in the past year, adapted from the Reproductive Autonomy coercion subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Kate E Doyle, Principal Investigator — Promundo-US; Ruti G Levtov, Principal Investigator — Prevention Collaborative; Fidele Rutayisire, Principal Investigator — Rwanda Men's Resource Centre; Shamsi Kazimbaya, Principal Investigator — Promundo-US; Felix Sayinzoga, Principal Investigator — Rwanda Biomedical Centre
Locations (1):
- Rwanda Men's Resource Centre, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doyle K, Levtov RG, Barker G, Bastian GG, Bingenheimer JB, Kazimbaya S, Nzabonimpa A, Pulerwitz J, Sayinzoga F, Sharma V, Shattuck D. Gender-transformative Bandebereho couples' intervention to promote male engagement in reproductive and maternal health and violence prevention in Rwanda: Findings from a randomized controlled trial. PLoS One. 2018 Apr 4;13(4):e0192756. doi: 10.1371/journal.pone.0192756. eCollection 2018. PMID 29617375
- [Derived] Doyle K, Levtov RG, Karamage E, Rakshit D, Kazimbaya S, Sayinzoga F, Sibomana H, Ngayaboshya S, Rutayisire F, Barker G. Long-term impacts of the Bandebereho programme on violence against women and children, maternal health-seeking, and couple relations in Rwanda: a six-year follow-up of a randomised controlled trial. EClinicalMedicine. 2023 Sep 26;64:102233. doi: 10.1016/j.eclinm.2023.102233. eCollection 2023 Oct. PMID 37781160